CLINICAL TRIAL: NCT02773290
Title: Phase 2/3 Study of Romiplostim(AMG531) in Subjects With Aplastic Anemia Refractory to or Ineligible for Immunosuppressive Therapy
Brief Title: Study of Romiplostim(AMG531) in Subjects With Aplastic Anemia
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Kyowa Kirin Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 531-002
Record Dates: First submitted 2016-05-09; First posted 2016-05-16 (Estimated); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: Aplastic Anemia
Keywords: Aplastic Anemia
MeSH Terms: conditions — Anemia, Aplastic | interventions — romiplostim

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Romiplostim (Experimental): Weekly Subcutaneous (SC) administration
  Interventions: Biological: Romiplostim

INTERVENTIONS:
Biological: Romiplostim — Weekly SC administration

SUMMARY:
The objective of this study is to evaluate the efficacy of romiplostim administered once weekly to Aplastic Anemia (AA) patients with thrombocytopenia refractory to or ineligible for immunosuppressive therapy in Japan and Korea.

Safety and pharmacokinetics of romiplostim after repeated administration will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Aplastic Anemia (AA) confirmed by peripheral blood and bone-marrow examinations, etc.
* Refractory to at least one course of immunosuppressive therapy including horse or rabbit anti-human thymocyte immunoglobulin (ATG); or ineligible for ATG treatment and refractory to cyclosporin (CyA)
* Thrombocytopenia defined as a platelet count of ≤ 30 × 10^9/L
* Preserving main organ function as a result of screening as follows;

  * Total bilirubin: < 1.5 times the upper limit of the laboratory normal range
  * Alanine aminotransferase: < 3.0 times the upper limit of the laboratory normal range
  * Aspartate aminotransferase: < 3.0 times the upper limit of the laboratory normal range
  * Creatinine value: ≤ 2.0 mg/dL
* An Eastern Cooperative Oncology Group performance status score of 0 to 2 at screening
* ≥ 20 years of age at the time of obtaining informed consent
* Patients who have provided written informed consent of their free will to participate in this study

Exclusion Criteria:

* Concurrent active infection not adequately responding to appropriate therapy
* Bone marrow reticulin grade of ≥ 2 based on the grading scale for reticulin indicated in Bone Marrow Pathology (2nd edition)
* Proportion of blasts in bone marrow > 2%
* Previous or concurrent active malignancies, other than localized tumors diagnosed more than one year previously and treated surgically with curative intent (basal cell carcinoma; or surgically resected in situ carcinoma of the cervix with an apparent success of ≥ 12 months prior to enrollment; as well as other cancers which have not been treated and remained disease-free for at least 5 years before enrollment are eligible)
* Clinically significant cardiac disease (class III or IV of the New York Heart Association classification; unstable angina pectoris; myocardial infarction within 6 months before enrollment; cardiac disease accompanied by angioplasty or stenting within 6 months before enrollment; or clinically significant cardiac arrhythmias) or uncontrollable hypertension
* Arterial or venous thrombosis within one year before enrollment
* Positive for anti-human immunodeficiency virus antibodies, hepatitis B surface antigen, or hepatitis C virus-RNA at screening
* Thrombocytopenia due to any other cause (e.g., myelodysplastic syndrome, idiopathic thrombocytopenic purpura, or liver cirrhosis)
* Patients with acute myeloblastic leukemia or chronic myelomonocytic leukemia
* Concurrent occurrence of hemolytic predominant paroxysmal nocturnal hemoglobinuria (Hemolytic predominant is defined as lactate dehydrogenase > 1.5 times the upper limit of the laboratory normal range)
* Uncontrolled diabetes mellitus
* Receiving other investigational products within 16 weeks before romiplostim treatment initiation
* Receiving any agent to treat AA, including the following agents before romiplostim treatment initiation;

  * ATG treatment within 6 months before romiplostim treatment initiation
  * CyA or anabolic steroid treatment within 6 weeks before romiplostim treatment initiation:

However, the patients who are treated with a CyA or anabolic steroid for at least 6 months before romiplostim treatment initiation may be enrolled if their blood cell count are stable at screening, and their dosage and administration will be kept for 6 weeks before romiplostim treatment initiation and during romiplostim dosing period.

* A history of polyethylene glycol-conjugated recombinant human megakaryocyte growth and development factor, recombinant human thrombopoietin (TPO), romiplostim, or other TPO-receptor agonists
* Having a plan to undergo hematopoietic stem cell transplantation within 1 year
* Having hypersensitivity to any recombinant protein E. coli derivative protein
* Lactating or pregnant women or women of child-bearing potential who have no intention of using oral contraceptives or birth control
* Having abnormalities by the cytogenetic test in bone marrow cells
* Patients who are considered to be ineligible for the study by the investigator or subinvestigator for reasons other than above

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2016-05; Primary Completion 2017-11-14 (Actual); Study Completion 2020-07-28 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects achieving a hematological response (any of the platelet response, erythroid response, and neutrophil response) at Week 27 | At 27 weeks after dosing

SECONDARY OUTCOMES:
Proportion of subjects with a hematological response at the end-of- treatment examination | Up to 52 weeks after dosing
Time from the first romiplostim administration to hematological response | Up to 52 weeks after dosing
In subjects receiving platelet transfusion as a pretreatment within 8 weeks prior to the first romiplostim administration; proportion of subjects with transfusion independence or decreased platelet transfusion requirement | Up to 52 weeks after dosing
Proportion of subjects achieving platelet response, erythroid response, or neutrophil response at each of Week 27 and end of treatment. | At 27 weeks and 52 weeks after dosing

CONTACTS AND LOCATIONS:
Locations (3):
- Japan (2):
  - Kanazawa
  - Tokyo
- Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jang JH, Mitani K, Tomiyama Y, Miyazaki K, Nagafuji K, Usuki K, Uoshima N, Fujisaki T, Kosugi H, Matsumura I, Sasaki K, Kizaki M, Sawa M, Hidaka M, Kobayashi N, Ichikawa S, Yonemura Y, Murotani K, Shimizu M, Matsuda A, Ozawa K, Nakao S, Lee JW. Predictive factors of romiplostim response in patients with refractory aplastic anemia: data from two clinical trials. Ann Hematol. 2025 Aug;104(8):4003-4011. doi: 10.1007/s00277-025-06337-7. Epub 2025 Jul 1. PMID 40593138